CLINICAL TRIAL: NCT01479595
Title: A Randomized Double-blind Multiple-dose Placebo-controlled Trial to Establish the Efficacy of QBX258 (Combination of VAK694 and QAX576) in Asthma That is Inadequately Controlled With Inhaled Corticosteroids and Long Acting Beta Agonists
Brief Title: A Study to Establish the Efficacy of QBX258 in Patients With Moderate to Severe Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQBX258X2201; 2011-003066-32 (EudraCT Number)
Record Dates: First submitted 2011-11-22; First posted 2011-11-24 (Estimated); Results first posted 2016-08-01 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-06

CONDITIONS: Asthma
Keywords: Asthma; Interleukin; QBX258; QAX576; VAK694
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- QBX258 (Experimental): Participants received QBX258 intravenous (iv) infusion every 4 weeks for up to 4 doses total.
  Interventions: Drug: QBX258
- Placebo (Placebo Comparator): Participants received placebo to QBX258 iv infusion every 4 weeks for up to 4 doses total.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QBX258 — QBX258 infusion, a combination of VAK694 and QAX576, was supplied to the Investigator as open label bulk medication. The planned dose of VAK694 (lyophilisate in vial, 150 mg/vial), was 3 mg/kg. The planned dose of QAX576 (lyophilisate in vial, 150 mg/vial), was 6 mg/kg.
  Arms: QBX258
Drug: Placebo — The placebo infusion was an equal volume of 5% dextrose for infusion and was provided by the clinical site.
  Arms: Placebo

SUMMARY:
This study is designed to investigate the efficacy and safety of QBX258 in subjects with moderate to severe asthma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with atopic asthma >1 year duration diagnosed according to the GINA guidelines.
* Subjects must weigh at least 50 kg to participate in the study, and must have a body mass index (BMI) within the range of 18 - 39 kg/m2.
* Asthma which is not adequately controlled on current treatment, as demonstrated by an Asthma Control Questionnaire (ACQ) score of > 1.5.
* FEV1 40 to 90% of predicted.

Exclusion Criteria:

* Diagnosed with COPD as defined by the GOLD guidelines
* Subjects who have had a respiratory tract infection within 4 weeks prior to screening.
* Women of child-bearing potential must use highly effective methods of contraception during dosing and for at least 18 weeks after last study drug administration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2012-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis Pharmaceuticals, Study Director — Novartis
Locations (19):
- United States (14):
  - Novartis Investigative Site, Anaheim, California
  - Novartis Investigative Site, Riverside, California
  - Novartis Investigative Site, Rolling Hills Estates, California
  - Novartis Investigative Site, San Marino, California
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Aventura, Florida
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Raleigh, North Carolina
  - Novartis Investigative Site, Winston-Salem, North Carolina
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Medford, Oregon
  - Novartis Investigative Site, Spartanburg, South Carolina
- Germany (3):
  - Novartis Investigative Site, Wiesbaden, Germany
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Frankfurt
- United Kingdom (2):
  - Novartis Investigative Site, London, United Kingdom
  - Novartis Investigative Site, Manchester

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were assigned to either QBX258 or placebo in a 2:1 ratio. Randomization was done by stratification of Q576R.
Period: Overall Study
Arm/Group | QBX258 | Placebo
Started | 44 | 21
PK Analysis Set | 42 | 0
Per Protocol Analysis Set | 41 | 20
Completed | 42 | 19
Not Completed | 2 | 2
Not completed — Protocol deviation | 0 | 1
Not completed — Adverse Event | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QBX258 | Placebo | Total
Number analyzed (Participants) | 44 | 21 | 65
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.5 (11.71) | 42.8 (13.54) | 42.6 (12.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 11 | 34
  Male | 21 | 10 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Asthma Control Questionnaire (ACQ) Score
Description: The ACQ consists of 7 questions assessing symptoms, rescue medication use and lung function. Except for lung function (FEV1), each question was scored on a 7-point scale where 0 = no impairment and 6 = maximum impairment. Scores ranged between 0 totally controlled to 6 (severely uncontrolled). Participants with a score below 1.0 are considered to have adequately controlled asthma. Participants with a score above 1.0 were considered not to be well controlled. A negative change from baseline indicates improvement.
Time Frame: Baseline and 12 weeks
Population: Participants from the per-protocol analysis set were considered for the analysis. Only participants who had both baseline and week 12 values were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | QBX258 | Placebo
Number analyzed (Participants) | 41 | 19
score on a scale | -0.513 (0.0970) | 0.001 (0.1487)
Statistical Analysis 1: Comparison: QBX258 vs Placebo; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis; Mean Difference (Net) = -0.514, 90% CI 2-sided [-0.811 to -0.217]

2. Secondary Outcome: Change in Forced Expiratory Volume in One Second (FEV1)
Description: FEV1 was assessed using central spirometry according to the American Thoracic Society/European Respiratory Society (ATS/ERS) guidelines.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QBX258 | Placebo
Number analyzed (Participants) | 41 | 19
Liters | 0.076 (0.0528) | 0.050 (0.0770)

3. Secondary Outcome: Change in Asthma Quality of Life Questionnaire (AQLQ) Score
Description: The AQLQ is a 32-item disease specific questionnaire designed to measure functional impairments that are most important to patients with asthma. It consists of 4 domains: symptoms, emotions., exposure to environmental stimuli and activity limitation.
  Patients were asked to recall their experiences during the previous 2 weeks and to score each item on a 7-point scale. The scale ranges from 1 to 7. The overall AQLQ score was the mean response to all 32 questions. Higher scores represent better outcomes.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | QBX258 | Placebo
Number analyzed (Participants) | 40 | 19
score on a scale | 0.580 (0.1294) | 0.468 (0.1878)

4. Secondary Outcome: Morning and Evening Peak Expiratory Flow (PEF) Rate
Description: Morning and evening PEFs were recorded on an electronic diary (e-diary). PEF was assessed twice daily approximately 12 hours apart and the measurements were recorded in the e-diary.
Time Frame: Baseline and 12 weeks
Population: No analysis was performed on the collected data with the eDiary device due to overall poor data quality (values were obtained that were not physiologically possible) and high variability. Therefore, there is no data to present for this outcome measure.
Arm/Group | QBX258 | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline in Maximum Expiratory Flow
Description: Maximum expiratory flow was assessed using central spirometry according to the American Thoracic Society/European Respiratory Society (ATS/ERS) guidelines.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/sec
Arm/Group | QBX258 | Placebo
Number analyzed (Participants) | 41 | 19
L/sec | 0.099 (0.4270) | 0.025 (0.3000)

6. Secondary Outcome: Number of Participants With Anti-QAX576 Antibodies or Anti-VAK694 Antibodies
Description: Anti-QAX576 and anti-VAK694 antibodies in serum were analyzed.
Time Frame: 12 weeks
Population: All randomized participants
Measure: Number; unit: Participants
Arm/Group | QBX258 | Placebo
Number analyzed (Participants) | 44 | 21
Participants | 2 | 2

7. Secondary Outcome: Observed Maximum Plasma Concentration Following Drug Administration at Steady State (Cmax,ss) of the QAX576 Analyte
Description: Blood samples were obtained to measure Cmax,ss.
Time Frame: days 1 (pre-dose and 2 hours post-dose), 15, 29 (pre-dose and 2 hours post-dose), 43, 57 (pre-dose and 2 hours post-dose), 71, 85 (pre-dose and 2 hours post-dose), 99, 113, 141, 183
Population: Participants from the per-protocol analysis set were considered for the analysis. Only participants who had week 12 values were included in the analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | QBX258
Number analyzed (Participants) | 40
ng/mL
  Q576R SNP stratum: QQ (n=21) | 169000 (47000)
  Q576R SNP stratum: RR/QR (n=19) | 184000 (85000)
  QBX258 (n=40) | 176000 (67300)

8. Secondary Outcome: Observed Maximum Plasma Concentration Following Drug Administration at Steady State (Cmax,ss) of the VAK694 Analyte
Description: Blood samples were obtained to measure Cmax,ss.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | QBX258
Number analyzed (Participants) | 40
ug/mL
  Q576R SNP stratum: QQ (n=21) | 56.7 (8.90)
  Q576R SNP stratum: RR/QR (n=19) | 58.6 (14.9)
  QBX258 (n=40) | 57.6 (12.0)

9. Secondary Outcome: Lowest Plasma Concentration Observed During a Dosing Interval at Steady State (Cmin,ss) of the QAX576 Analyte
Description: Blood samples were obtained to measure Cmin,ss.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | QBX258
Number analyzed (Participants) | 40
ng/mL
  Q576R SNP stratum: QQ (n=21) | 37500 (11900)
  Q576R SNP stratum: RR/QR (n=19) | 32200 (9930)
  QBX258 (n=40) | 35000 (11200)

10. Secondary Outcome: Lowest Plasma Concentration Observed During a Dosing Interval at Steady State (Cmin,ss) of the VAK694 Analyte
Description: Blood samples were obtained to measure Cmin,ss.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | QBX258
Number analyzed (Participants) | 40
ug/mL
  Q576R SNP stratum: QQ (n=21) | 10.7 (2.69)
  Q576R SNP stratum: RR/QR (n=19) | 9.83 (2.94)
  QBX258 (n=40) | 10.3 (2.81)

11. Secondary Outcome: Change From Baseline in Fractional Exhaled Nitric Oxide (FeNO)
Description: FeNO was assessed as a measure of airway inflammation. An FeNO machine was used to obtain the FeNO measurements. FeNO measurements were obtained prior to the spirometry assessments.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: parts per billion (ppb)
Arm/Group | QBX258 | Placebo
Number analyzed (Participants) | 36 | 15
parts per billion (ppb) | -3.67 (3.580) | 2.21 (5.393)

ADVERSE EVENTS:
Arm/Group | QBX258 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/44 | 1/21
Other Adverse Events (participants affected / at risk) | 13/44 | 7/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QBX258 (N=44) | Placebo (N=21)
ABORTION (Pregnancy, puerperium and perinatal conditions) | 0 | 1
LARYNGEAL OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QBX258 (N=44) | Placebo (N=21)
NAUSEA (Gastrointestinal disorders) | 3 | 0
VOMITING (Gastrointestinal disorders) | 3 | 0
NASOPHARYNGITIS (Infections and infestations) | 4 | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 2
HEADACHE (Nervous system disorders) | 5 | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.